CLINICAL TRIAL: NCT05670054
Title: Cyclin Dependant Kinase 4/6 (CDK4/6) Inhibitors as a Second Line Treatment in Metastatic Breast Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Manar Hamed, assistant lecturer medical oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.22.07.674
Record Dates: First submitted 2022-12-17; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — Quality of Life; Progression-Free Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- palbociclib + fulvestrant (Active Comparator): Arm A includes patients who receive palbociclib 125 mg tab/day for 3 weeks and 1 week rest+ Fulvestrant 500 mg IM injection d1, d15, d29 1st cycle then every month
  Interventions: Drug: comparing both arms as regard the objective response rate, toxicity profile, quality of life, progression free survival
- Ribociclib + fulvestrant (Active Comparator): Arm B includes patients who receive ribociclib 200 mg 3 tabs/day for 3 weeks and 1 week rest+ Fulvestrant 500 mg IM injection d1, d15, d29 1st cycle then every month
  Interventions: Drug: comparing both arms as regard the objective response rate, toxicity profile, quality of life, progression free survival

INTERVENTIONS:
Drug: comparing both arms as regard the objective response rate, toxicity profile, quality of life, progression free survival — comparing both arms as regard the objective response rate, toxicity profile, quality of life, progression free survival

SUMMARY:
Breast cancer is the commonest malignancy among females and one of the leading causes of death worldwide. Many drugs have been developed over the years to try to extend survival among these patients including cyclin dependant kinase inhibitors. Cyclin dependant kinase inhibitors (CDK inhibitors) mainly Palbociclib (PAL), ribociclib (RIB) and abemaciclib (ABM) are approved for treatment of hormone receptor positive, HER2 negative advanced breast cancer in the 1st line and subsequent lines in combination with aromatase inhibitors or fulvestrant. Studies showed that they extend progression free survival and recently they showed overall survival benefit. In this study investigators compare Palbociclib+ fulvestrant VS Ribociclib + fulvestrant as a second line treatment in metastatic ER+ve her2 -ve BC in oncology center mansoura university egyptian patients.

DETAILED DESCRIPTION:
Breast cancer is the commonest malignancy among females and one of the leading causes of death worldwide. Many drugs have been developed over the years to try to extend survival among these patients including cyclin dependant kinase inhibitors. Cyclin dependant kinase inhibitors (CDK inhibitors) mainly Palbociclib (PAL), ribociclib (RIB) and abemaciclib (ABM) are approved for treatment of hormone receptor positive, HER2 negative advanced breast cancer in the 1st line and subsequent lines in combination with aromatase inhibitors or fulvestrant. Studies showed that they extend progression free survival and recently they showed overall survival benefit. In this study investigators compare Palbociclib+ fulvestrant VS Ribociclib + fulvestrant as a second line treatment in metastatic ER+ve her2 -ve BC in oncology center mansoura university egyptian patients. The efficacy and comparative toxicity of CDK inhibitors were indirectly compared in a number of trials. Despite differences in inclusion criteria and follow-up length, second-line trials showed similar characteristics.

Unfortunately, despite the similar efficacy and overall response rate (ORR) and a slightly different but near-identical spectrum of adverse events, both agents have not been directly compared with each other. This study aims to fill that gap, and evaluate the toxicity, tolerability and response rate of ribociclib plus fulvestrant versus palbociclib plus fulvestrant, to inform the decision makers.

ELIGIBILITY:
Inclusion Criteria:

* - Pathologically proven diagnosis of adenocarcinoma of the breast with evidence of metastatic disease either progression on adjuvant hormonal or progression on 1st line hormonal for metastatic disease.
* Documentation of ER-positive and/or PR-positive and HER2 negative.
* Prior use of endocrine therapy.
* age >18 years old.
* ECOG: 0-2
* Postmenopausal is defined as: age>60 years old or < 60 years old with cessation off menstruation for at least 12 months and FSH or E2 in postmenopausal range or patients who underwent bilateral oophorectomy.
* Premenopausal is defined if not meeting the criteria of postmenopausal. They are obligated to receive LHRH agonist with their treatment.

Exclusion Criteria:

* - Age < 18 years old
* Patients with advanced/metastatic, symptomatic, visceral spread(visceral crisis) , that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions [pleural, pericardial, peritoneal], pulmonary lymphangitis, and over 50% liver involvement).
* 2nd malignancy other than breast cancer
* ECOG more than 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The rate of objective response and clinical benefit | the last patient recruited in the study will be followed up for at least 6 months
  compare objective response rate and clinical benefit rate between the 2 arms
Incidence and grade of toxicity | the last patient recruited in the study will be followed up for at least 6 months
  compare the incidence and grade of toxicity between the 2 arms
Compare Quality of life score of the patients using EORTC core quality of life questionaire version C-30 | each patient will answer the QOL score at D0, 3rd and 6 months of treatment as long as he is hasn't progressed on treatment during the 1st 6 months
  compare the level of deterioration of the quality of life score between the 2 arms

CONTACTS AND LOCATIONS:
Overall Officials: manar hamed, MD, Principal Investigator — Oncology center mansoura university
Locations (1):
- Oncology center mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the results of the study will be shared and published
Supporting Information: Study Protocol, SAP
Time Frame: at january 2023 for 3 years
Access Criteria: All data will be available to the fellow researchers